CLINICAL TRIAL: NCT04104516
Title: A Brief Messaging Lifestyle Modification Program for Patients With Non-small Cell Lung Cancer
Brief Title: Lifestyle Modification Program for Lung Cancer Patients - Physical Activity Preference
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant Professor, The University of Hong Kong
Other Study IDs: UW19-597-1
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: Lifestyle modification; Lung Cancer; Preferences
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is the leading cause of deaths in the world. Engagement in physical activity can provide important benefits for cancer patients. The current study is a cross-sectional questionnaire survey and in-depth interview to understand the physical activity preferences of patients with lung cancer. This process could help to develop a lifestyle modification program based on our patients' needs and preferences.

DETAILED DESCRIPTION:
Lung cancer is one of the most common cancer globally and locally. Patients with lung cancer are in a uniquely difficult situation in their disease, comorbidities, and treatment that may lead to worsened symptoms and many negative health consequences, including fatigue, irritability, and impaired daytime functioning.

Physical activity (PA) is defined as 'any bodily movement produced by skeletal muscle that results in energy expenditure'. Several health benefits of increased PA have been reported for people with cancer. PA plays a critical role across the cancer trajectory, from prevention through to post-diagnosis and has been proposed as an alternative for improving physical and psychosocial health outcomes, reducing cancer recurrence, and cancer-specific and all-cause mortality. However, most of the findings were predominantly in breast and colorectal cancers. The PA dosage required to attain health benefits across these cancer groups is not uniform, nor is it clear whether the results can be applied to other groups of people with cancer.

The current study includes a cross-sectional questionnaire survey and an in-depth interview. It aims to understand the current physical activity practice and preference of patients with lung cancer, which could help to develop a lifestyle modification program based on our patients' needs and preferences.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above;
* Diagnosis with non-small cell lung cancer
* General condition stable, either is undergoing or finished treatment
* Able to speak and read Chinese
* Able to complete the self-administered questionnaire
* Mental, cognitive and physically fit for joining the trial as determined by the clinician or responsible investigator

Exclusion Criteria:

* Mentally unfit for answering questionnaire
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Preference on physical activity program | immediately after obtaining written consent
  Outcome-based questions with categorical choices

SECONDARY OUTCOMES:
Current physical activity practise | immediately after obtaining written consent
  Outcome-based questions with categorical choices
Preference on information to be received | immediately after obtaining written consent
  Outcome-based questions with categorical choices

CONTACTS AND LOCATIONS:
Overall Officials: LAI YK Agnes, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The patient consent did not include sharing personal information to other researchers

REFERENCES:
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Background] Peddle-McIntyre CJ, Singh F, Thomas R, Newton RU, Galvao DA, Cavalheri V. Exercise training for advanced lung cancer. Cochrane Database Syst Rev. 2019 Feb 11;2(2):CD012685. doi: 10.1002/14651858.CD012685.pub2. PMID 30741408
- [Derived] Lai AYK, Choi A, Yiu DYS, Sun Y, Kwok TTO, Yeung WF, Lam DCL, Lam TH. Digital health and physical activity: Insights from advanced lung cancer patients in Hong Kong. Asia Pac J Oncol Nurs. 2025 Jul 19;12:100759. doi: 10.1016/j.apjon.2025.100759. eCollection 2025 Dec. PMID 40831612
- See also: World health Organisation - Cancer — https://www.who.int/news-room/fact-sheets/detail/cancer